CLINICAL TRIAL: NCT06199167
Title: The Effect of Action Observation Therapy on Upper Extremity Function in Children With Obstetric Brachial Plexus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve Çalışkan, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MÇalışkan
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Brachial Plexus Palsy; Obstetric; Injury
Keywords: Obstetric Brachial Plexus Injury; Action Observation Therapy; Upper Limb Function; Visual Motor Imagination
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants did not know the other intervention and were not exposed to each other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy (Experimental): The Action Observation Therapy group watched each ADL activity for two minutes through pre-prepared videos and then repeated the movement they watched for three minutes.
  Interventions: Behavioral: Action Observation Therapy
- Photo Observation (Experimental): The Photo Observation group observed the photographs taken from the video for two minutes and then practised the movement described for three minutes.
  Interventions: Behavioral: Photo Observation

INTERVENTIONS:
Behavioral: Action Observation Therapy — The Action Observation Therapy group watched each ADL activity for two minutes through pre-prepared videos and then repeated the movement they watched for three minutes. In the 15-session treatment, a total of 18 ADL activities.
  Arms: Action Observation Therapy
Behavioral: Photo Observation — The Photo Observation group observed the photographs taken from the video for two minutes and then practised the movement described for three minutes. In the 15-session treatment, a total of 18 ADL activities.
  Arms: Photo Observation

SUMMARY:
Introduction: Musculoskeletal problems in the upper limb (UL) caused by nerve damage following Obstetric Brachial Plexus Injury (OBPI) and disorders affecting the use of the UL can limit activities of daily living (ADLs) and limit the child's participation in school and society. Method: Twenty-six children with OBPY aged between 6-17 years participated in the study and were randomised AOT and Photo Observation (PO) groups in equal numbers by stratified randomisation. In the 15-session treatment, a total of 18 ADL activities related to personal care, dressing, eating and preparation, transfer and mobilisation activities, reaching, and sports activities were studied with six exercises per session. The AOT group watched each ADL activity for two minutes through pre-prepared videos and then repeated the movement they watched for three minutes. The PO group observed the photographs taken from the video for two minutes and then practised the movement described for three minutes. The same sequence was continued for six exercises and one session was completed in approximately 30 minutes. Abilhand-Kids (AK), Seated Medicine Ball Throw (SMBT), Modified Push-up Test (MPT), Functional Reach Test (FRT), Lateral Reach Test (LRT), Brachial Plexus Outcome Measurement (BPOM), Gilbert and Raimondi Score (GRS), Box Block Test (BBT) were performed before and after the treatment.

DETAILED DESCRIPTION:
Introduction: Musculoskeletal problems in the upper limb (UL) caused by nerve damage following Obstetric Brachial Plexus Injury (OBPI) and disorders affecting the use of the UL can limit activities of daily living (ADLs) and limit the child's participation in school and society. No study investigating the effect of EGT in children with OBPY has been found in the literature. Based on this deficiency, we aimed to investigate the effect of EGT in children with OBPY in a randomised controlled study.

Hypotheses of our study H0: There is no difference between Action Observation Therapy and Photo Observation in improving upper extremity functional skills in children with OBPY.

H1: There is a difference between Action Observation Therapy and Photo Observation in improving upper extremity functional skills in children with OBPY.

Method: Twenty-six children with OBPY aged between 6-17 years participated in the study and were randomised AOT and Photo Observation (PO) groups in equal numbers by stratified randomisation. In the 15-session treatment, a total of 18 ADL activities related to personal care, dressing, eating and preparation, transfer and mobilisation activities, reaching, and sports activities were studied with six exercises per session. The AOT group watched each ADL activity for two minutes through pre-prepared videos and then repeated the movement they watched for three minutes. The PO group observed the photographs taken from the video for two minutes and then practised the movement described for three minutes. The same sequence was continued for six exercises and one session was completed in approximately 30 minutes. Abilhand-Kids (AK), Seated Medicine Ball Throw (SMBT), Modified Push-up Test (MPT), Functional Reach Test (FRT), Lateral Reach Test (LRT), Brachial Plexus Outcome Measurement (BPOM), Gilbert and Raimondi Score (GRS), Box Block Test (BBT) were performed before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6-18
* OBPY diagnosed in Type 1, Type 2a, Type 2b group according to Narakas classification system
* Triceps brachii muscle strength above 3/5 in manual muscle strength assessment
* Family and child agree to take part in the study

Exclusion Criteria:

* History of upper extremity surgery and Botox in the last 6 months
* Difficulty in understanding the commands given
* Visual and hearing problems
* Finding of shoulder dislocation
* Orthopaedic problems associated with OBPY

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Abilhand Kids | 5 weeks
  ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved
Seated Medicine Ball Throw | 5 weeks
  This test measures upper body (arm) strength and explosive power. By keeping the back in contact with the wall the strength of the arms only are tested.
Modified Push-up Test | 5 weeks
  The Modified Push-Up Test is used to measure upper body strength endurance and trunk stability. This variation, which uses a modified technique with a clap behind the back while in the 'down' position and a touch from one hand to the other in the 'up' position.
Functional Reach Test | 5 weeks
  Functional Reach Test (FRT) is the maximal distance one can reach forward beyond arm's length while maintaining a fixed standing position.
Lateral Reach Test | 5 weeks
  The LR Test measures postural stability in the medial-lateral direction by assessing the maximum distance an individual can reach laterally beyond arm's length at shoulder height, while maintaining a fixed base of support in the standing position

SECONDARY OUTCOMES:
Brachial Plexus Outcome Measurement | 5 weeks
  The Brachial Plexus Outcome Measure (BPOM) scale was developed in 2012 by Emily S. Ho and contains 14 items that measure activity and self-evaluation.
Gilbert and Raimondi Score | 5 weeks
  The Gilbert and Raimondi Assessment System is an assessment system developed by Gilbert to assess shoulder and elbow function and Raimondi to assess hand function.
Box Block Test | 5 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. The BBT is composed of a wooden box divided in two compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No